CLINICAL TRIAL: NCT04274309
Title: Evaluation of the Medical Device ex Vivo ENDOSWIR in Patient Operated for a Tonsillectomy : a Preliminary Cohort Study Proof of Concept (ENDOSWIR-AMYG)
Brief Title: Safety Validation of EndoSWIR Device
Acronym: ENDO-AMYG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Institut National de la Santé et de la Recherche Médicale, Institute for Advanced Biosciences (Unknown); Commissariat A L'energie Atomique (Other Government); Lynred (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC19.388; 2019-A03333-54 (Other: ID RCB)
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Optical Guided Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient's tissues exposed: Tonsil of each patient will be imaged using the medical device
  Interventions: Device: EndoSWIR
- Patient's tissues not exposed: Tonsil of each patient will not be imaged using the medical device
  Interventions: Device: EndoSWIR

INTERVENTIONS:
Device: EndoSWIR — Exposition of the respected tissues to the camera

SUMMARY:
Head and neck cancer has an incidence of 600,000 cases per year worldwide (6th among cancers) and cause 380,000 death per year. Surgical resection is guided by the surgeon's inspection and palpation of the tumor. The prognosis of patients depends on the quality of the lesion's resection. The ENDOSWIR dispositive developed by engineers of Atomic Energy Comity of Grenoble allows for reliable and accurate analysis of tumor margins.

The camera provides a spectral analysis of the tissues according to their composition. We want to show that the prognosis of patients is improved by the use of this device. For that we need to prove first that it is not toxic for tissue analysis.

DETAILED DESCRIPTION:
ENDOSWIR dispositive is a InGaAs (Indium Gallium Arsenide) camera working at ambient temperature. The light is a quartz-tungstene-halogeno (QTH) source and the collected beam is filtered to illuminate in different precise wavelength bands in the short wave domain.

We will use it on tonsil tissue just after tonsillectomy and just before the histological analysis.

ELIGIBILITY:
Inclusion Criteria:

* Tonsillectomy

Exclusion Criteria:

* suspicion of Head-and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men or Women more than 18
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Tissue integrity | 1 day
  Histological score : evaluation of cellular cohesion and denaturation of epithelial cells and conjunctive support tissue

CONTACTS AND LOCATIONS:
Overall Officials: Christian RIGHINI, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No